CLINICAL TRIAL: NCT01871454
Title: Effect of Pentoxifylline and Vitamin E in Preventing Radiation-induced Toxicity in the Treatment of Recurrent or New Primary NSCLC Using Stereotactic Ablative Radiotherapy in Patients Previously Treated With Thoracic Radiation
Brief Title: Safety of Pentoxifylline and Vitamin E With Stereotactic Ablative Radiotherapy (SABR) in Non-small Cell Lung Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Neal Edward Dunlap, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-RAD-13-Pentoxifylline
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancers
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy (SABR) plus pentoxifylline (Experimental): standard of care radiotherapy (SABR) plus pentoxifylline and Vitamin E
  Interventions: Radiation: stereotactic ablative radiotherapy (SABR); Drug: Pentoxifylline

INTERVENTIONS:
Radiation: stereotactic ablative radiotherapy (SABR) — standard of care radiation therapy
Drug: Pentoxifylline — pentoxifylline

SUMMARY:
The objective of this prospective phase II protocol is to assess the toxicity and efficacy of pentoxifylline and SABR in the re-treatment of recurrent or new lung cancers

ELIGIBILITY:
3.1 Inclusion Criteria: - Eligibility Criteria

3.1.1 Age >/= 18 years

3.1.2 ECOG performance status 0-1 3.1.3 Histologically proven diagnosis of a prior thoracic malignancy treated with thoracic external beam radiotherapy with or without systemic chemotherapy

3.1.4 Pathologic or clinical diagnosis of a new or loco-regional recurrent lung malignancy. A reasonable attempt should be made to make a pathologic diagnosis of malignancy (ie. bronchoscopy, CT guided lung biopsy)

* Loco-regional is defined as recurrence within the region of the primary tumor or adjacent draining lymph node regions.
* The new lesion or loco-regional recurrence must be within or adjacent to the previously irradiated treatment volume.

3.1.5 Imaging as follows:

* CT scan of the chest with IV contrast within 8 weeks of registration
* Whole body PET scan within 8 weeks of registration

3.1.6 Pulmonary function test (PFTs), including diffusion capacity within 8 weeks of registration

3.1.7 Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential.

3.1.6 Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control

3.1.7 Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

- 3.2 Exclusion Criteria

3.2.1. No previously reported thoracic radiotherapy

3.2.2. FEV1 <20% predicted and/or DLCO <20% predicted

3.2.2. Pregnant women or lactating women

3.2.3 Chemotherapy within 4 weeks of the initiation of SABR

3.2.4 Plans to administer systemic chemotherapy overlapping with radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
primary endpoint is to estimate overall treatment-related toxicity | 36 months-end of trial

SECONDARY OUTCOMES:
Estimate progression free survival | 12 months
Estimate tumor failure | 12 months
estimate overall survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Neal E Dunlap, MD, Principal Investigator — James Graham Brown Cancer Center-U of Louisville
Locations (1):
- James Graham Brown Cancer Center, U of Louisville, Louisville, Kentucky, United States